CLINICAL TRIAL: NCT04574882
Title: Using Digital Data to Predict Cardiovascular Health and Health Care Utilization
Brief Title: Using Digital Data to Predict CHD
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833699
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases
Keywords: digital data; digital health
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients ages 30-74 with and without CHD (IICD 10: I63, I20-I25 ) within the last 5 years.
  Interventions: Other: Survey
- Control: Patients aged 30-74 who have non-cardiovascular-related history
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Interested participants may complete the informed consent online. After informed consent, the participant will be asked to share the digital data types that they use (Facebook, Instagram, Twitter, Google search, step data) and then participants will complete a cross-sectional survey.

SUMMARY:
This project seeks to identify and characterize features derived from digital data (e.g. social media, online search, mobile media) which are associated with coronary heart disease (CHD) and related risk factors, and develop models that use digital data and conventional predictive models to predict CHD risk and health care utilization.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in the US. While secondary prevention approaches have improved longevity of patients, risk factors and adverse health behaviors (e.g., physical inactivity, smoking) are highly prevalent, and in most contemporary series, less than 1% of adults meet all factors of ideal CV health. The logistics and practicalities of meeting the goal of ideal CV health have not been clearly elucidated. Practice guidelines recommend using the Framingham risk score (FRS) or other risk prediction tools to classify patients' risk of CV disease. These models however are imprecise and there is increasing focus on identifying markers that provide better measures of risk. As digital platforms are increasingly used to document lifestyle and health behaviors, data from digital sources may provide a window into manifestations of novel risk factors and potentially a better characterization of existing risk factors. While it seems like a cliche to mention the profound impact of digital data on everyday lives, there is indeed great substance in the opportunities these new media provide for understanding behavioral, social, and environmental determinants of health. This project seeks to identify and characterize features derived from digital data (e.g. social media, online search, mobile media) which are associated with coronary heart disease (CHD) and related risk factors, and develop models that use digital data and conventional predictive models to predict CHD risk and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 74 years of age
* Willing to sign informed consent
* Primarily English speaking (for language analysis)
* Has an account on any of the following digital data platforms (Facebook, Instagram, Twitter Reddit, Google (gmail), or smartphone or wearable device such as Apple Health, Fitbit, Samsung Health, MapMyFitness or Garmin) and willing to share data
* If has social media account, Instagram or Facebook, willing to share historical and prospective data (60 days) If has Google (gmail) account, willing to download and share google takeout zip file
* If has smartphone or wearable device, willing to share step data
* Willing to share access to medical health records
* Willing to share healthcare insurance information

Exclusion Criteria:

* Patient does not meet age inclusion criteria above
* Does not use and post on digital data sources we are studying or unwilling to donate data
* Patient is in severe distress, e.g. respiratory, physical, or emotional distress
* Patient is intoxicated, unconscious, or unable to appropriately respond to questions

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will identify patients ages 30-74 with and without CHD (ICD 9:414.0, ICD 10: I63, I20-I25)
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Case | Control
Started | 326 | 455
Completed | 194 | 333
Not Completed | 132 | 122

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case | Control | Total
Number analyzed (Participants) | 326 | 455 | 781
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.5) | 59.5 (9.2) | 60.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were allowed to select 'Prefer not to say' for their sex. 38 case and 43 control participants selected that option
  Participants
    number analyzed (Participants) | 288 | 412 | 700
    Female | 141 | 287 | 428
    Male | 147 | 125 | 272
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 10 | 13 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 152 | 207
  White | 217 | 254 | 471
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 43 | 35 | 78

OUTCOME MEASURES:

1. Primary Outcome: Latent Dirichlet Allocation (LDA) Topics - Topics / Themes Discussed Between Patients With and Without Heart Disease
Description: The primary outcome is topics and features (derived using the LDA method for clustering language data).
  For each participant, we included all available Facebook wall posts from the start of their account history through data collection, regardless of whether they occurred before or after a CHD diagnosis. We examined associations between linguistic features (unigrams, LIWC categories, LDA topics) and cardiovascular case status (CHD presence vs absence) using Pearson correlation and logistic regression. Latent LDA, a systematic method to identify text-based themes, was applied to generate 200 clusters of co-occurring words ("topics"). For each feature type (unigram, LIWC category, LDA topic), we fit separate logistic regression models and calculated Pearson correlation coefficients to assess predictive value for case status. Each language-derived feature was encoded as a normalized frequency count per user to enable consistent comparison across participants.
Time Frame: Through study completion, an average of 3 years
Population: To evaluate predictive performance for ASCVD risk, we used regression and classification analyses. Pearson correlations assessed how language features predicted continuous risk scores. For classification, we measured AUC for binary risk (≥10% vs <10%) and standard risk categories. Three logistic regression models were tested: language alone, demographics alone, and combined. Arms/groups were combined because the goal was to predict ASCVD risk continuously and categorically across participants.
Measure: Number (100% Confidence Interval); unit: proportion probability AUC (Area Under t
Groups:
- Binary Classification (≥10% vs. <10%) Binary Classification; All Risk Categories: To evaluate predictive performance for atherosclerotic cardiovascular disease (ASCVD) risk scores, we conducted both regression and classification analyses. Pearson correlation coefficients were used to measure how well language features predicted continuous ASCVD risk scores. For classification tasks, we assessed the area under the receiver operating characteristic curve (AUC) for models predicting both binary risk status (high versus low ASCVD risk, defined as ≥10% versus <10%) and established ASCVD risk categories (<5%, 5%-7.4%, 7.5%-9.9%, and ≥10%).
Arm/Group | Binary Classification (≥10% vs. <10%) Binary Classification | All Risk Categories
Number analyzed (Participants) | 119 | 219
proportion probability AUC (Area Under t
  Demographics only | 0.85 [0 to 1] | 0.87 [0 to 1]
  LIWC only | 0.55 [0 to 1] | 0.67 [0 to 1]
  Unigrams only | 0.61 [0 to 1] | 0.71 [0 to 1]
  LDA only | 0.64 [0 to 1] | 0.67 [0 to 1]
  LIWC + Demographics (age, sex, race) | 0.79 [0 to 1] | 0.80 [0 to 1]
  Unigrams + Demographics (age, sex, race) | 0.61 [0 to 1] | 0.74 [0 to 1]
  LDA + Demographics (age, sex, race) | 0.81 [0 to 1] | 0.82 [0 to 1]

2. Other Pre Specified Outcome: CHD Event
Description: Reliability in predicting CHD related event in patient as measured by Framingham Risk Score.
  The Framingham Risk Score (FRS) is a validated means of predicting cardiovascular disease (CVD) risk. Input variables include age, cigarette smoking, total cholesterol, HDL cholesterol, systolic blood pressure measurement and treatment for hypertension. Point values are calculated based on each of these risks. A 10-year risk score can be derived as a percentage. Risk scores range from 0-20%.
  Low Risk: Less than 10% risk that you will develop a heart attack or die from coronary disease in the next 10 years.
  Intermediate risk: A 10 to 20% risk that you will develop a heart attack or die from coronary disease in the next 10 years.
  High Risk: A greater than 20% risk that you will develop a heart attack or die from coronary disease in the next 10 years.
Time Frame: Through study completion, an average of 3 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Health Care Utilization
Description: Prediction of cost for health care utilization between heart disease and non- heart disease subjects measured by insurance claims data
Time Frame: Through study completion, an average of 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: This study was cross-sectional and no adverse event data was collected.
Description: This study was cross-sectional and no adverse event data was collected. Due to this study design feature the number of participants at risk for Serious Adverse Events is zero, the number of participants at risk for All-Cause Mortality is zero, and the number of participants at risk for Other (Not Including Serious) Adverse Events is zero.
Arm/Group | Case | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04574882/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04574882/SAP_002.pdf